CLINICAL TRIAL: NCT04532515
Title: Seal-G and Seal-G MIST Study for Reinforcement and Protection of Colonic Anastomoses in Subjects Undergoing Colonic Resection
Brief Title: Seal-G / Seal-G MIST Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: ClinSearch (Other); Advanced Medical Solutions Israel (Sealantis) Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DLG-072-06
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Colon Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Seal-G Product Family variants will be used as the study device (Treatment) according to the following scheme:
  1. Seal-G Surgical Sealant [Seal-G]- will be applied on colonic anastomosis created by extra-corporal approach.
  2. Seal-G MIST System [Seal-G MIST]- will be applied on colonic anastomosis created by intra-corporal approach.
  Intended Use: Seal-G/Seal-G MIST are surgical sealants intended for use as an adjunct to standard closure techniques for reinforcement and protection of gastrointestinal anastomoses.
  Device is an adjunct device and will be applied following standard colon resection surgery and creation of primary anastomosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seal G / Seal-G MIST (Experimental): Seal-G Surgical Sealant [Seal-G]- will be applied on colonic anastomosis created by extra-corporal approach.
  Seal-G MIST System [Seal-G MIST]- will be applied on colonic anastomosis created by intra-corporal approach.
  Interventions: Device: Seal-G Surgical Sealant; Device: Seal-G MIST System

INTERVENTIONS:
Device: Seal-G Surgical Sealant — Seal-G is a surgical sealant intended for use as an adjunct to standard closure techniques for reinforcement and protection of gastrointestinal anastomoses.
  Device is an adjunct device and will be applied following standard colon resection surgery and creation of primary anastomosis
  Other Names: Seal-G
Device: Seal-G MIST System — Seal-G MIST is a surgical sealant intended for use as an adjunct to standard closure techniques for reinforcement and protection of gastrointestinal anastomoses.
  Device is an adjunct device and will be applied following standard colon resection surgery and creation of primary anastomosis
  Other Names: Seal-G MIST

SUMMARY:
A prospective, multi-center, open label, study to evaluate safety and performance of Seal-G and Seal-G MIST in reinforcing colonic anastomosis, in subjects undergoing Colon Resection surgery

DETAILED DESCRIPTION:
Seal-G and Seal-G MIST Surgical Sealants are intended for the reinforcement and protection of gastrointestinal anastomosis. The Seal-G and Seal-G MIST devices share the same Alginate based sealant technology and intended purpose. The devices only differ in their method of application, The Seal-G device is designed for spread application by extra-corporal approach, and the Seal-G MIST device is designed for spray application by intra-corporal approach.

The proposed Clinical Investigation aims to collect clinical evidence on the devices' usage, including safety, performance and usability.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs and dates a written ICF, indicates an understanding of the study procedures and follow-up requirements and is willing to comply with them.
2. Subject is aged 18 years to 80 years
3. Subject is scheduled for elective open or laparoscopic (including robotic) colon cancer resection surgery with primary anastomosis (excluding low anterior resection)

Exclusion Criteria:

1. Anastomosis is expected to be ≤ 10cm from anal verge
2. Surgery involves stoma creation
3. Subject who underwent a prior pelvic radiation therapy
4. Subject with a BMI > 40 or <19
5. Subject with ASA status higher than 3
6. Albumin level < 3 gr/dl
7. Total bilirubin >1.5 mg/dL
8. Hemoglobin level < 8mg/dl on day of surgery
9. Subject has a diagnosis of bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, and carcinomatosis
10. Subject treated with immunosuppressive agents within 28 days prior to study enrollment (including corticosteroids)
11. Serious or uncontrolled co-existent diseases (e.g. severe cardiovascular disease, congestive heart failure, recent myocardial infarction within 6 months from surgery, significant vascular disease, active or uncontrolled autoimmune disease, active or uncontrolled infection, uncontrolled DM with episodes of hospitalization due to hypo or hyperglycemia within 6 months of surgery)
12. Subject known to have distant metastases, such as liver, lung, bone etc. metastases (not including local and regional lymph nodes)
13. Subject with known sensitivity to Indigo carmine dye (FD&C 2/ E132)
14. Subject who according to the investigator clinical judgement is not suitable for participation in the study or is at risk
15. Subject requires more than one anastomosis during the surgery
16. Subject is scheduled for another surgery during the follow up period of this study
17. Subjects who cannot comply with study visits/ procedures or have poor compliance (e.g. mentally handicapped, prisoners, etc.)

Intraoperative Exclusion Criteria:

Subjects who meet any of the following intra-operative exclusion criteria will be considered as screen failures and will not be eligible for the study:

1. Positive leak test requires anastomosis takedown and/or re-anastomosis.
2. Additional resection (not including tissue biopsy) of non-colonic solid organ (e.g. Liver resection, uterus, bladder, seminal vesicle, ureter)
3. Subjects whom anastomosis is ≤10 cm from the anal verge
4. Subject received intraoperative sealant, glue or any buttressing material for the study related anastomosis, other than the Seal-G/Seal-G MIST
5. Subject received two or more units of PC transfusion during surgery
6. Subject has peritoneal carcinomatosis or any other metastasis observed by the surgeon

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of surgeries with full sealant coverage - successful application | At time of surgery
  1- The surgeon applied the sealant over the full circumference of the anastomosis (successful application).
  0 - The surgeon did not fully cover the anastomosis circumference

SECONDARY OUTCOMES:
Proportion of subjects with clinical anastomotic leaks | Up to 30 days post-surgery
  1 - The subject had a clinical anastomotic leak 0 - The subject did not have a clinical anastomotic leak
Proportion of subjects with subclinical / radiological leaks | Up to 30 days post-surgery
  1 - The subject had a Subclinical /radiological anastomotic leak 0 - The subject did not have a Subclinical /radiological anastomotic leak
Proportion of subjects with at least one Serious Adverse Event | Up to 30 days post-surgery
  1 - The subject had any Serious adverse event 0 - The subject did not have Serious adverse event
Proportion of subjects that had a reoperation | Up to 30 days post-surgery
  1 - The subject had any event of reoperation 0 - The subject did not have reoperation
Hospital length of stay | Up to 30 days post-surgery
  Measured by the time for "Ready to be discharged" (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Kamar, MD, Study Director — Advanced Medical Solutions Israel (Sealantis) Ltd.
Locations (2):
- Israel (2):
  - Sheba Medical Center (Tel Hashomer), Ramat Gan
  - Shamir (Assaf Harofeh) Medical Center, Rishon LeZiyyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamar M, Kanani F, Spinelli A, Jayne D, Segev L, Tutton M, Montroni I, Tulchinsky H, Shimonov M, Lavy R, Zmora O. Efficacy and safety of novel alginate-based sealants (SEAL-G and SEAL-G MIST) in reducing anastomotic leakage following colorectal anastomosis: a prospective multicenter study. Ann Coloproctol. 2025 Oct;41(5):424-433. doi: 10.3393/ac.2025.00297.0042. Epub 2025 Oct 23. PMID 41125251